CLINICAL TRIAL: NCT04100538
Title: Fibromyalgia: Impacts of Different Phenotypes on Quality of Life and the Effects of Technology-assisted and Tailored Health Coaching
Brief Title: Quality of Life and the Effects of Tailored Health Coaching in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Pei-Shan, Tsai, Bio-Behavior Research Laboratory, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N201809035
Record Dates: First submitted 2019-09-09; First posted 2019-09-24 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Fibromyalgia
Keywords: Health coaching; Quality of Life
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive the technology-assisted program by health coach twice a week during the 10-week treatment period. The health coach will be an experienced master-prepared nurse who has extensive and in-depth knowledge about fibromyalgia and has previously worked in direct contact with patients with fibromyalgia in a research project.
  Interventions: Behavioral: health coach
- control group (No Intervention): The control group will receive technology-assisted informational support twice a week during the 10-week treatment period. Each technology-assisted informational support will last for approximately 10-30 min consisting of 15-min questions-and-answers regarding the educational materials and 15-min debriefing.

INTERVENTIONS:
Behavioral: health coach — The health-coaching program includes (1) my file, (2) lesson, (3) self-assessment, and (4) interaction modules. My file allows participants recording their disease history. The lesson includes knowledge of fibromyalgia, stress and relaxation, emotion and positive thinking, sleep hygiene, communication skills, and exercise. The self-assessments includes symptom diary, exercise and general diary. The interaction encourages participants interacting with peers and the health coach. Participants can share practical advices, strategies, real-life examples or questions via texts or photos in "share garden". Participants can connect to the health coach via "contact with health coach". The coach will provide comments or responses approximately 10-30 min for each time. The coach will monitor each participant's lesson list and attendance for each lesson. The health coach will also guide the participants to create their own tailored programs according to participants' predominant symptom subtypes.
  Arms: Intervention group

SUMMARY:
Specific Aims:

1. To identify phenotypes of patients with fibromyalgia according to symptom clusters and to compare differences in quality of life (QOL) among different phenotypes.
2. To examine the effects of technology-assisted and tailored health coaching in comparison to telephone support on health status, QOL, pain catastrophizing, and self-efficacy in patients with fibromyalgia.

Methods:

For Aims 1, the investigators will conduct a cross-sectional study and enroll 300 patients with fibromyalgia. Symptoms will be assessed using the Numerical Rating Scale, Athens Insomnia Scale, Functional Assessment of Cancer Therapy cognition scale, Beck Depression Index-II, Beck Anxiety Index, and Fatigue Severity Scale. The World Health Organization Quality of Life-Brief Form (WHOQOL-BREF) questionnaire will be used to assess participants' overall QOL. Hierarchical cluster analyses will be used to identify fibromyalgia phenotypes according to pain, physical, and psychological variables. A series of multivariate analysis of variance analyses will be used to compare the differences in WHOQOL-BREF scores among those phenotypes.

For Aims 2, the investigators conduct an assessor-blind, parallel-group, randomized controlled trial and enroll 110 participants with fibromyalgia. Participants will be randomized to a health coaching group and a control group. The tailored, interactive health-coaching program will be delivered via mobile applications during a 10-week training period. The control group will receive standard education materials and weekly telephone support. The primary outcomes are the revised Fibromyalgia Impact Questionnaire and WHOQOL-BREF scores; the secondary outcomes are pain catastrophizing score and self-efficacy, which will be examined at baseline, post-training, and the 3th month follow-up. Data will be analyzed according to the intention-to-treat principle. To determine the effectiveness of health coaching on primary and secondary outcomes, differences in outcome variables will be analyzed with mixed-effects linear regression models. The between-group differences at the two posttests examined using a mixed-model will include group x time interaction. The investigators will adjust for the baseline score on the outcome variable and for demographics and comorbidities that differ significantly between the intervention and control groups at baseline.

DETAILED DESCRIPTION:
Background:

Fibromyalgia is a chronic pain syndrome predominantly affecting adult women. It is characterized by widespread musculoskeletal pain accompanied by physical and psychological symptoms, such as sleep disturbance, cognitive impairment, fatigue, stiffness, anxiety, and depression. The complexity and heterogeneity of clinical symptoms have been observed among patients with fibromyalgia. Variability in the intensity of fibromyalgia-related symptoms differentially impact patients' degree of disability, quality of life, and pain. Several cluster studies have sought to identify clinically relevant phenotypes based on disease symptoms.

However, those studies only focused on selected physical and psychological symptoms to construct the symptom clusters. Few studies included cognitive variables into the clusters and few studies investigated the difference in the quality of life (QOL) and functional status among different subgroups or phenotypes of patients with fibromyalgia. Therefore, identification of phenotypes based on a comprehensive set of symptoms and determining differential impacts of fibromyalgia phenotypes on quality of life among patients with fibromyalgia is important, both scientifically and clinically as this information may help the healthcare professionals select appropriate treatments.

Recent meta-analyses showed that multicomponent treatments are effective in reducing pain and improving QOL in patients with fibromyalgia, probably owing to the complexity of pain and heterogeneity of symptoms. Pain catastrophizing and self-efficacy are powerful predictors for disability. Therefore, an effective program must include tailored, multicomponent therapy for decreasing catastrophizing and increasing self-efficacy, which in turn may improve symptoms, functional status, and quality of life.

Specific aims of the study are:

1. To identify phenotypes of patients with fibromyalgia according to symptom clusters and to compare differences in QOL among different phenotypes.
2. To examine the effects of technology-assisted and tailored health coaching in comparison to telephone support on health status, QOL, pain catastrophizing, and self-efficacy in patients with fibromyalgia.

Methods

Specific Aim 1-Study 1 (Year 1-2):

Participants will be recruited via referrals from the physicians and from the community by on-line advertisements posted on websites or social media, and advertisement (posters and flyers) posted in public places. Based on Formann's method, which states that the maximum number of clustering variables should be m, where sample size = 2^m, the number of clustering variables was limited to 7. A recent study identified three fibromyalgia subgroups among 345 participants. Therefore the investigators will enroll 300 participants for Study 1.

Specific Aim 2 - Study 2 (Year 1-3):

Similarly to Study 1, participants will be recruited via referrals from the physicians and from the community by on-line advertisements posted on websites or social media, and advertisement (posters and flyers) posted in public places. Naturally, subjects who are screened for eligibility for participation in Study 1 will be offered a chance to participate in Study 2. The sample size is estimated based on the expected treatment effect size for the primary outcome. The treatment effect size of non-pharmacological treatments for improving QOL in fibromyalgia patients was 0.73 according to results from a previous meta-analysis study. Assuming a type I error of 0.05, a type II error of 0.2 and an effect size of 0.73, 44 subjects per group will achieve a 0.8 power with a 2-sided test according to the results of the power analysis. 110 participants will be enrolled to accommodate planned subgroup analyses and to allow for a 25% dropout rate.

Randomization sequence generation and concealment:

After obtaining written consent and completion of baseline measurements, eligible participants will be randomly assigned in a 1:1 ratio with the use of permuted blocks of ten each to an intervention group (n = 55) and a control group (n = 55). An independent research assistant who will not involve in participant recruitment, enrollment, and data collection will generate randomization sequence using computerized software. The generated random sequence will be concealed in sequentially numbered, opaque envelopes until the participant is assigned. Appropriate random allocation and allocation sequence concealment will reduce selection bias.

Blinding:

To minimize detection bias, assigning an independent research assistant who is masked to the group assignment for baseline and post-test data collections will ensure assessor blindness.

Study procedures and data collections:

The study protocol describing the flow of participants into the intervention and control groups and data collections in different study weeks is depicted in Figure 1. Briefly, subjects respond to advertisements or referred by physicians will undergo screening for eligibility. After confirming the eligibility and obtaining written informed consent, participants will complete the baseline assessment of demographic variables, medical history, lifestyles variables, primary outcomes and secondary outcomes. Participants will then be assigned to the study groups according to the pre-generated randomization sequence. Both groups will repeat the assessment of the primary and secondary outcomes immediately after the 10 weeks of training period (posttest 1) and at the 3-month follow-up (posttest 2).

Statistical analyses:

Differences in baseline data will be determined using the Mann-Whitney U-tests, chi-square tests, and t-tests for independent samples. Comparisons of group means at baseline, and the two post-tests will be performed for normally distributed primary and secondary outcomes using independent t test. Effect size (Cohen's d) will be calculated for each outcome variable. To determine the effectiveness of technology-assisted health coaching on primary and secondary outcomes, differences in outcome variables will be analyzed with mixed-effects linear regression models with the covariance structure unstructured. The investigators will perform statistical analyses according to the intention-to-treat principle. All missing vales will be imputed using the last value carry-forward method. The between-group differences at the two post-test assessments will be examined using a mixed-model in which group and time interaction will be included. The investigators will adjust for the baseline score on the outcome variable and for demographics and comorbidities that differ significantly between the health coaching group and control group at baseline.

ELIGIBILITY:
Study1.

Inclusion Criteria:

1. 20 years of age and older.
2. A Polysymptomatic Distress Scale (PDS) score of 13 and greater.

Exclusion Criteria: No

Study2.

Inclusion Criteria:

1. 20 years of age and older.
2. A Polysymptomatic Distress Scale (PDS) score of 13 and greater.
3. Capable of using web-application via smartphone.

Exclusion Criteria:

1. Medical history of significant head injury or neurological disorder.
2. Malignant neoplasm.
3. Women with pregnancy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2022-11-06 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQR) at baseline | baseline
  The FIQR is an instrument that assesses the current health status of patients with fibromyalgia in clinical and research settings; it comprised three domains: physical function, overall effect of fibromyalgia, and fibromyalgia symptoms (pain, fatigue, un refreshing sleep, stiffness, anxiety, depression, tenderness to touch, memory, balance and environmental sensitivity). All 21 questions are graded on a 0-10 numeric scale (no difficulty to very difficult); higher FIQR score indicates greater symptom severity. The reliability coefficients ranged from 0.56 on the pain score to 0.95 for physical function. A Chinese version of the FIQR will be used.
Fibromyalgia Impact Questionnaire (FIQR) after the 10 weeks of training period | after the 10 weeks of training period
  The FIQR is an instrument that assesses the current health status of patients with fibromyalgia in clinical and research settings; it comprised three domains: physical function, overall effect of fibromyalgia, and fibromyalgia symptoms (pain, fatigue, un refreshing sleep, stiffness, anxiety, depression, tenderness to touch, memory, balance and environmental sensitivity). All 21 questions are graded on a 0-10 numeric scale (no difficulty to very difficult); higher FIQR score indicates greater symptom severity. The reliability coefficients ranged from 0.56 on the pain score to 0.95 for physical function. A Chinese version of the FIQR will be used.
Fibromyalgia Impact Questionnaire (FIQR) at 3 months postintervention | 3 months postintervention
  The FIQR is an instrument that assesses the current health status of patients with fibromyalgia in clinical and research settings; it comprised three domains: physical function, overall effect of fibromyalgia, and fibromyalgia symptoms (pain, fatigue, un refreshing sleep, stiffness, anxiety, depression, tenderness to touch, memory, balance and environmental sensitivity). All 21 questions are graded on a 0-10 numeric scale (no difficulty to very difficult); higher FIQR score indicates greater symptom severity. The reliability coefficients ranged from 0.56 on the pain score to 0.95 for physical function. A Chinese version of the FIQR will be used.
World Health Organization Quality of Life - BREF (WHOQOL-BREF) at baseline | baseline
  This study will use the WHOQOL-BREF to determine participants' overall QOL. The WHOQOL-BREF was developed by World Health Organization (WHO)76, which is a brief self-report instrument to measure subjects' overall quality of life. The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale. The Taiwan version of WHOQOL-BREF which contains 28 items has a Cronbach's α for internal consistency of 0.70 to 0.77.
World Health Organization Quality of Life - BREF (WHOQOL-BREF) after the 10 weeks of training period | after the 10 weeks of training period
  This study will use the WHOQOL-BREF to determine participants' overall QOL. The WHOQOL-BREF was developed by World Health Organization (WHO)76, which is a brief self-report instrument to measure subjects' overall quality of life. The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale. The Taiwan version of WHOQOL-BREF which contains 28 items has a Cronbach's α for internal consistency of 0.70 to 0.77.
World Health Organization Quality of Life - BREF (WHOQOL-BREF) at 3 months postintervention | 3 months postintervention
  This study will use the WHOQOL-BREF to determine participants' overall QOL. The WHOQOL-BREF was developed by World Health Organization (WHO)76, which is a brief self-report instrument to measure subjects' overall quality of life. The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale. The Taiwan version of WHOQOL-BREF which contains 28 items has a Cronbach's α for internal consistency of 0.70 to 0.77.

SECONDARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | baseline,after the 10 weeks of training period (posttest 1), and at 3 months postintervention (posttest 2)
  The Beck Depression Inventory-II (BDI-II), a scale designed to assess depression symptom severity, will be used to assess depressive symptoms in this study. The BDI II is a self-administered 21-item questionnaire in which responses are ranked from 0 to 3, with greater scores corresponding to more frequent symptoms. The BDI-II has high internal consistency (α = 0.91), and an average test-retest reliability of 0.72 across 20 studies. The BDI-II scores range between 0 and 63, with increasing scores indicating more severe ratings of depression. BDI-II yields reliable, internally consistent and valid scores in a primary care medical setting. A Chinese version of the BDI-II will be used.
Beck Anxiety Inventory (BAI) | baseline, after the 10 weeks of training period (posttest 1), and at 3 months postintervention (posttest 2)
  The Beck Anxiety Inventory (BAI)-Chinese version, a 21-question multiple-choice self-report questionnaire will be used for measuring the severity of anxiety. The BAI is a 4-point Likert-type rating scale that measures a person's feeling of being bothered by his/her symptoms in the past week (0 = not bothered at all, 3 = almost unbearable). Each item is descriptive of subjective, somatic, or panic-related symptoms of anxiety. The BAI has a maximum score of 63 with higher scores representing higher levels of anxiety. Previous research results have supported its reliability and validity. A Chinese version of the BAI will be used.
Pain Catastrophizing Scale (PCS) | baseline, after the 10 weeks of training period (posttest 1), and at 3 months postintervention (posttest 2)
  The PCS is a self-administered questionnaire consisting of 13 items that assess negative emotional and cognitive processes (e.g., helplessness, rumination, pessimism, and magnification of symptoms) will be used to evaluate pain catastrophizing. The PCS uses a 5-point scale to measure the frequency with which individuals experience pain-related thoughts and feelings. Participants are asked to indicate the degree to which they have certain thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale; a total score is yielded (ranging from 0-52), along with three subscale scores assessing rumination, magnification and helplessness. The PCS has been shown to have adequate to excellent internal consistency and concurrent validity82. A validated Chinese version of the PCS will be used.
Pain Self-Efficacy Questionnaire (PSEQ) | baseline, after the 10 weeks of training period (posttest 1), and at 3 months postintervention (posttest 2)
  The PSEQ is a 10-item self-report inventory that assesses the strength and generality of a patient's self-efficacy beliefs and his or her confidence to accomplish a range of activities in the presence of chronic pain. Patients are asked to rate how confident they are at that time despite the presence of their pain in performing ten activities listed by selecting a number on a 7 point scale, where 0 equals ''not at all confident'' and 6 equals ''completely confident''. Scores on the PSEQ may range from 0 to 60, with higher scores indicating stronger self-efficacy beliefs. The Cronbach's α for internal consistency is 0.9285. A validated Chinese version of the PSEQ will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Shan Tsai, PhD, Study Chair — Taipei Medical University
Locations (1):
- Bio-Behavior Research Laboratory, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No